CLINICAL TRIAL: NCT05971225
Title: Prospective Multicenter Observation Study on the Association Between Remote Monitoring and Clinical Outcome in Heart Failure Patients (Verifying Remote Monitoring Effect on Net Cardiovascular Outcome; RemoteVerify (RêVe))
Brief Title: Verifying Remote Monitoring Effect on Net Cardiovascular Outcome; RemoteVerify (RêVe)
Acronym: ReVe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Vincent's Hospital, Korea (Other)
Collaborators: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RemoteVerify
Record Dates: First submitted 2023-07-13; First posted 2023-08-02 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Congestive Heart Failure; Defibrillators; Cardiac Resynchronization Therapy
Keywords: remote monitoring; congestive heart failure; Defibrillators; cardiac resynchronization therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: one group with experience of in-office device monitoring >6 months the other group without experience of in-office device monitoring
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Follow up group (Active Comparator): participants with experience of >6 months in-office device interrogation, then started remote monitoring
  Interventions: Other: remote monitoring only
- Remote group (Experimental): participants with newly implanted device with study agreement, and then started remote monitoring
  Interventions: Other: remote monitoring only

INTERVENTIONS:
Other: remote monitoring only — remote monitoring only can replace in-office device monitoring
  Other Names: in office monitoring

SUMMARY:
This study investigates the impact and safety of wireless monitoring on the prognosis of heart failure patients with implanted pacemakers and defibrillators. It aims to examine the frequency of unplanned early hospital visits and the early diagnosis/intervention of disease exacerbation based on the presence or absence of wireless monitoring. Additionally, the study analyzes the influence of wireless monitoring on the patient's disease progression as well as satisfaction of the study participants.

ELIGIBILITY:
Inclusion Criteria:

* consented heart failure patients (LVEF<=40%) with Biotronik wireless monitoring capable ICD/CRTs aged >20 years
* patients who are new to remote monitoring

Exclusion Criteria:

* For patients with a life expectancy of less than 6 months. If patient do not understand the contents of wireless monitoring or it is difficult to fill out the consent form due to cognitive decline.

If wireless monitoring is performed with a patient enrolled in another clinical trial which remote monitoring may affect the previous enrolled study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Unplanned early visits for cardiac causes1 (Patient) | 6 months
  i. Unplanned hospitalization/admission due to patient's condition changes -> Patients' needs-driven early visits
Unplanned early visits for cardiac causes2 (Patient) | 12months
  i. Unplanned hospitalization/admission due to patient's condition changes -> Patients' needs-driven early visits
Unplanned early visits for cardiac causes3 (Patient) | 18months
  i. Unplanned hospitalization/admission due to patient's condition changes -> Patients' needs-driven early visits
Unplanned early visits for cardiac causes4 (Patient) | 24months
  i. Unplanned hospitalization/admission due to patient's condition changes -> Patients' needs-driven early visits
Unplanned early visits for cardiac causes1 (Clinic) | 6months
  ii. Hospitalization/Admission due to alerts on the implanted cardiac device following wireless monitoring -> Clinician-driven early visits
Unplanned early visits for cardiac causes2 (Clinic) | 12months
  ii. Hospitalization/Admission due to alerts on the implanted cardiac device following wireless monitoring -> Clinician-driven early visits
Unplanned early visits for cardiac causes3 (Clinic) | 18months
  ii. Hospitalization/Admission due to alerts on the implanted cardiac device following wireless monitoring -> Clinician-driven early visits
Unplanned early visits for cardiac causes4 (Clinic) | 24months
  ii. Hospitalization/Admission due to alerts on the implanted cardiac device following wireless monitoring -> Clinician-driven early visits

SECONDARY OUTCOMES:
Acute myocardial infarction (heart attack) or cerebrovascular events (stroke) | 6,12,18,24 months
  ACS, CVA
Thromboembolic events (such as pulmonary embolism) | 6,12,18,24 months
  Systemic thromboembolic events
Worsening of heart failure leading to hospitalization | 6,12,18,24 months
  HF related admission
Cardiac-related deaths | 6,12,18,24 months
  Cardiac cause deaths
Overall mortality | 6,12,18,24 months
  overall deaths

CONTACTS AND LOCATIONS:
Locations (1):
- St. Vincent's Hospital, Suwon, Kyonggi Do, South Korea

IPD SHARING:
Plan to Share IPD: No
It will not be open because its sensitive data, however, if there's reasonable request, data can be acquired after de-identification of the participants.